CLINICAL TRIAL: NCT06424262
Title: A Pivotal, Prospective, Multi-centre, Randomised Controlled, 6-month Blinded Investigation Followed by a 6-month Open-label Phase Evaluating the Efficacy of a Dexamethasone Eluting Slim Straight Electrode (CI622D) in the Reduction of Impedance as Compared to a Standard Slim Straight Electrode (CI622) in a Newly Implanted Adult Population With Post-linguistic, Bilateral, Moderately Severe to Profound Sensorineural Hearing Loss.
Brief Title: Performance and Hearing-related Outcomes in Adults Implanted With the CI622D Dexamethasone-eluting Cochlear Implant Compared to Those Implanted With a Standard Cochlear Implant (CI622)
Acronym: DETECT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Collaborators: QbD Clinical (Industry); Avania (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLTD5815
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-03

CONDITIONS: Hearing Loss, Bilateral Sensorineural; Hearing Loss, Sensorineural; Hearing Loss, Bilateral; Hearing Loss, Cochlear
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Sensorineural; Hearing Loss, Bilateral

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CI622D (Experimental): Investigational Medical Device (IMD)
  Interventions: Device: CI622D
- CI622 (Active Comparator): An approved medical device
  Interventions: Device: CI622

INTERVENTIONS:
Device: CI622D — A dexamethasone-eluting Slim Straight electrode
  Arms: CI622D
Device: CI622 — A standard Slim Straight electrode
  Arms: CI622

SUMMARY:
This clinical study will test a newly developed cochlear implant known as CI622D. This experimental cochlear implant has been designed to slowly release a drug called dexamethasone. Dexamethasone works to ease inflammation, which is common after any surgical procedure. The goal is to learn if there are added benefits in implant performance and hearing outcomes with the dexamethasone-releasing cochlear implant (CI622D) vs. the standard cochlear implant (CI622) without dexamethasone. The study will be conducted in adults with sensorineural hearing loss, a type of hearing loss caused by damage to the inner ear or auditory nerve. The study participants will undergo a series of tests that include testing their implant and their hearing. They will also complete questionnaires to see how they rate their hearing ability and their overall general health.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older (at time of consent)
* Clinically established post-linguistic bilateral moderately severe to profound sensorineural hearing loss
* Meets local candidacy criteria for cochlear implantation
* Compromised functional hearing with a hearing aid in the ear to be implanted
* Willing to participate in and comply with all requirements of the protocol, including willingness to be randomised to either arm
* Evidence of pneumococcal vaccination (e.g., Pneumovax) according to local guidelines prior to randomisation
* Candidate is proficient in the language used to assess speech perception performance
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Planned for a partial insertion of the electrode array
* Intra-axial (within the brain) lesions or deafness due to lesions of the acoustic nerve affecting the ear to be implanted
* Middle ear infection (including acute otitis media, chronic otitis media, suppurative otitis media, or serous drainage) in the ear to be implanted either at the time of surgery or within 3 months prior to enrolment
* Active autoimmune disease or active immunosuppressive therapy
* Any of the following in the ear to be implanted within 3 months prior to enrolment: history of prior otologic surgery including grommets, or tympanic membrane perforation
* Previously reported diagnosis of auditory neuropathy, in the ear to be implanted
* Previously reported diagnosis, in the ear to be implanted, of Large Vestibular Aqueduct Syndrome (LVAS), Meniere's disease, or cochlear hydrops
* Ossification, otosclerosis, malformation or any other cochlear anomaly, such as common cavity, that might prevent complete insertion of the electrode array, as confirmed by imaging, in the ear to be implanted
* Current cerebrospinal fluid (CSF) shunts or drains, existing perilymph fistula, temporo- parietal skull fracture or CSF leaks
* History of bacterial meningitis
* Known allergic reaction or contraindication to dexamethasone or corticosteroids
* Severe, or poorer, bilateral sensorineural hearing loss prior to 5 years of age, as reported by the subject
* Severe, or poorer, sensorineural hearing loss of more than 20 years, as reported by the subject, in the ear to be implanted
* Prior cochlear implantation, in either ear
* Medical plan for cochlear implantation during the clinical investigation, contralateral to the ear to be implanted
* Medical or psychological conditions that contraindicate general anaesthesia, surgery or participation in the clinical investigation, as determined by the investigator
* Women who are pregnant
* Unrealistic expectations on the part of the subject, regarding the possible benefits, risks, and limitations that are inherent to the surgical procedure(s) and prosthetic devices as determined by the Investigator
* Additional disabilities that may affect the subject's participation or safety during the clinical investigation, as determined by the Investigator
* Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator
* Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as spouse, parent, child, or sibling to the study candidate
* Cochlear employees or employees of Contract Research Organisations or contractors engaged by Cochlear for the purposes of this investigation
* Current participation, or participation in another interventional clinical study/trial in the past 30 days, involving an investigational drug or device (unless Cochlear sponsored and determined by investigator or Sponsor to not impact this investigation)
* Subjects recruited at a French site who are not affiliated with social security
* Subjects recruited at a French site who are under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Difference in the mean monopolar 1+2 (MP1+2) impedance between CI622D (Investigational Medical Device) and CI622 (control device) at 6 months post-activation | 6 months post-activation
  The impedance will be measured across the active electrodes of the implant for each participant.

SECONDARY OUTCOMES:
Difference in mean (within-subject) change in word recognition score in the preferred unilateral listening mode in quiet from pre-implantation to post-activation with CI622D compared with CI622 | Pre-implantation, 3, 6, 12 months post-activation
  Change in word recognition score will be measured from pre-implantation to 3, 6 and 12 months post-activation.
Proportion of participants who experience an adverse event and the proportion of participants who experience a device deficiency with CI622D and CI622 | Throughout study (12 months)
  Adverse events will be recorded as overall, by severity, by relatedness to device or procedure, or by seriousness. Device deficiency will be recorded as overall and by type.
Difference in the mean unaided acoustic hearing thresholds pre-operatively, and from activation to post-activation between CI622D and CI622 | Pre-operative, 0, 3, 6, 12 months post-activation
  Unaided acoustic hearing thresholds will be measured pre-operatively, at activation, and 3, 6 and 12 months post-activation.
Mean within-subject change in word recognition score in the preferred unilateral listening mode in quiet from pre-implantation to post-activation with CI622D | Pre-implantation, 3, 6, 12 months post-activation
  Word recognition scores will be measured at pre-implantation and 3, 6 and 12 months post-activation.
Mean change (within-subject) in word recognition score in the preferred bilateral listening mode in quiet from pre-implantation to post-activation with CI622D | Pre-implantation, 3, 6, 12 months post-activation
  Word recognition scores will be measured at pre-implantation and 3, 6 and 12 months post-activation.
Difference in mean (within-subject) change in word recognition score in the preferred bilateral listening mode in quiet from pre-implantation to post-activation with CI622D compared with CI622 | Pre-implantation, 3, 6, 12 months post-activation
  Change in word recognition score will be measured from pre-implantation to 3, 6 and 12 months post-activation.
Difference in mean (within-subject) change in sentence recognition score in noise in the preferred unilateral listening mode from pre-implantation to post-implantation with CI622D compared with CI622 | Pre-implantation, 3, 6, 12 months post-activation
  Change in sentence recognition score (Matrix test + 10 SNR) will be measured from pre-implantation to 3, 6 and 12 months post-activation.
Difference in mean (within-subject) change in sentence recognition score in noise in the preferred bilateral listening mode from pre-implantation to post-implantation with CI622D compared with CI622 | Pre-implantation, 3, 6, 12 months post-activation
  Change in sentence recognition score (Matrix test + 10 SNR) will be measured from pre-implantation to 3, 6 and 12 months post-activation.
Difference in the mean nested bipolar impedances and MP1+2 impedances between CI622D and CI622 measured intraoperatively and from activation to post-activation | Intraoperative, at activation and 3, 6 and 12 months post-activation.
  Nested bipolar impedances will be measured intraoperatively, at activation and 3, 6 and 12 months post-activation. MP1+2 impedances will be measured intraoperatively, at activation and 3 and 12 months post-activation
Difference in the mean estimated sound processor battery life for CI622D compared from activation to post-activation with CI622 | 0, 3, 6,12 months post-activation
  The estimated sound processor battery life (hours per day) will be measured at activation, 3, 6, and 12 months-post activation.
Difference in mean within-subject changes in global score on the Speech, Spatial, and Qualities of Hearing Scale (SSQ12) from pre-implantation to post-activation between CI622D and CI622 | Pre-implantation, 3, 6, 12 months post-activation
  Global SSQ12 scores will be measured at pre-implantation and 3, 6 and 12 months post-activation.
Difference in mean within-subject changes in global Health Utilities Index III (HUI3) from pre-implantation to post-activation between CI622D and CI622 | Pre-implantation, 3, 6, 12 months post-activation
  Global HUI3 scores will be measured at pre-implantation and 3, 6 and 12 months post-activation.

CONTACTS AND LOCATIONS:
Overall Officials: Antje Aschendorff, Principal Investigator — Universitätsklinikum Freiburg
Locations (11):
- Australia (5):
  - Macquarie University, Sydney, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Westmead Private Hospital, Sydney, New South Wales
  - St Vincent Private Hospital, Melbourne, Victoria
  - Royal Victorian Eye and Ear Hospital, Melbourne E., Victoria
- France (3):
  - Centre Hospitalier Universitaire de Lille, Lille
  - Hôpital Universitaire Pitié-Salpêtrière, Paris
  - Centre Hospitalier Universitaire Toulouse, Toulouse
- Germany (2):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Freiburg Im Breisgau
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
- Manchester Royal Infirmary, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No